CLINICAL TRIAL: NCT01490255
Title: Comparison of the Pharmacodynamic Effects of RanOlazine Versus aMlodipine on Platelet Reactivity in Stable Patients With Coronary Artery Disease Treated With Dual ANtiplatelet Therapy - The ROMAN Randomized Study
Brief Title: Pharmacodynamic Effects of Ranolazine Versus Amlodipine on Platelet Reactivity
Acronym: ROMAN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 654/2011/D
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
Keywords: platelet reactivity; aspirin; clopidogrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ranolazine; Amlodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Active Comparator): Patients will receive ranolazine (750 mg bid) for 15 days
  Interventions: Drug: Ranolazine
- Amlodipine (Active Comparator): Patients will receive amlodipine (10 mg once daily) for 15 days
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Ranolazine — os, 750 mg, twice per day, for 15 days
  Other Names: Ranexa®, Gilead, USA
  Arms: Ranolazine
Drug: Amlodipine — os, 10 mg, once daily, 15 days
  Other Names: Norvasc®, Pfizer, USA
  Arms: Amlodipine

SUMMARY:
No previous study has assessed the potential of ranolazine to interfere with levels of platelet reactivity in patients with coronary artery disease who are treated with dual antiplatelet therapy.

Aim of this study is to compare the pharmacodynamic effects of maintenance doses of ranolazine versus amlodipine on platelet reactivity in patients with coronary artery disease who are treated with dual antiplatelet therapy.

DETAILED DESCRIPTION:
Patients with coronary artery disease (CAD) are often treated with dual antiplatelet therapy (DAT), including aspirin and clopidogrel, to prevent from recurrent atherothrombotic events.

Levels of platelet reactivity in patients on DAT can be influenced by concomitant treatment with medications that inhibit the CYP3A4 system involved in the activation of clopidogrel, such as calcium channel blockers, potentially interfering with its clinical benefits. Importantly, calcium channel blockers, such as amlodipine, are commonly used for relief of ischemic symptoms in patients with CAD.

Ranolazine is a novel antianginal drug that reduces intracellular sodium and calcium accumulation and constitutes a pharmacologic alternative to calcium channel blockade.

However, no previous study has assessed the potential of ranolazine to interfere with levels of platelet reactivity in CAD patients on DAT.

The primary objective of this study is to compare the pharmacodynamic effects of maintenance doses of ranolazine versus amlodipine on platelet reactivity in patients with CAD on DAT.

ELIGIBILITY:
Inclusion Criteria:

* Angiographically-proven coronary artery disease
* Class I indication to dual antiplatelet therapy because of recent (<12 months) percutaneous coronary intervention and/or recent acute coronary syndrome (<12 months)
* Stable clinical conditions
* Able to understand and willing to sign the informed consent form

Exclusion Criteria:

* Use of other drug interfering with CYP activity such as proton pump inhibitors
* Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of platelet reaction units | After 15 days of treatment with each drug
  Absolute changes in platelet reactivity (expressed as P2Y(12) reaction units by the point-of-care VerifyNow assay [Accumetrics, San Diego, California])

SECONDARY OUTCOMES:
Frequency of high platelet reactivity | After 15 days of treatment with each drug
  Frequency of high platelet reactivity with the two study treatments (as defined by a Platelet Reaction Unit value>240

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pelliccia, MD, Principal Investigator — University La Sapienza, Rome, IT
Locations (2):
- Italy (2):
  - San Raffaele Pisana, Rome
  - University La Sapienza, Rome